CLINICAL TRIAL: NCT01446705
Title: Evaluation of VLER_Indiana Health Information Exchange Demonstration Project
Brief Title: Evaluation of VLER-Indiana Health Information Exchange Demonstration Project
Acronym: VLER-IHIE
Status: Completed | Type: Observational
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: Regenstrief Institute, Inc. (Other)
Responsible Party: Sponsor
Other Study IDs: IIR 11-058
Record Dates: First submitted 2011-04-27; First posted 2011-10-05 (Estimated); Results first posted 2016-01-29 (Estimated); Last update posted 2019-05-16 (Actual); Status verified 2019-05

CONDITIONS: Diabetes Mellitus; Asthma; Cardiovascular Diseases; Heart Failure; Osteoporosis
MeSH Terms: conditions — Diabetes Mellitus; Asthma; Cardiovascular Diseases; Heart Failure; Osteoporosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- No Exchange: Patients in this arm will represent Veterans seen at the Indianapolis VA Medical Center (VAMC) for whom information exchange has not been activated.
  Interventions: Other: Non-Active Health Information exchange
- Enrolled in Exchange: Patients in this arm will represent Veterans seen at the Indianapolis VAMC for whom information exchange has been activated by the patient choosing to "opt-in."
  Interventions: Other: Active Health Information Exchange

INTERVENTIONS:
Other: Active Health Information Exchange — Patients selected to share data between the VA & external healthcare agencies.
  Groups: Enrolled in Exchange
Other: Non-Active Health Information exchange — Patients not selecting to share data
  Groups: No Exchange

SUMMARY:
Three out of four Veterans receive a portion of their care from non-VA providers. On April 9, 2009, President Barack Obama directed the Department of Veterans Affairs and the Department of Defense to create the Virtual Lifetime Electronic Record (VLER). On August 2010, Secretary of Veterans Affairs Eric K. Shinseki visited Indianapolis, and after visiting with leaders from the VA Health Services Research & Development (HSR&D) Center of Excellence and the Regenstrief Institute, he made the following public comments regarding the latest partnership between the two institutions: "This new technology allows safer, more secure, and private access to electronic health information which, in turn, enhances our ability to continue providing Veterans with the quality care that they have earned."

This new technology refers to the VLER HEALTH program that the Indianapolis VA is now implementing in partnership with the Regenstrief Institute and Indiana Health Information Exchange (IHIE). This VA-IHIE demonstration project is intended to create the capacity for VA institutions to exchange health information with community partners.

Investigators from the VA HSR&D Center on Implementing Evidence-Based Practice are active collaborators in building and implementing this program. The VA-IHIE program provides the bi-directional exchange of health information between VA and non-VA providers. Based on our pilot study of linked VA-IHIE data, investigators are conducting an evaluation of the impact of the VA-IHIE demonstration project upon health care quality and cost of Veterans by taking advantage of the initiation of the implementation as a natural experiment.

DETAILED DESCRIPTION:
This study will perform a pre-post evaluation of the VA-IHIE implementation, with a concurrent control group, among Veterans seen at the Indianapolis VA. Data on care received by Veterans will be obtained for one year before, and one year after, VA-IHIE enrollment. Patients will be recruited into the VA-IHIE program in a rolling manner over the course of a year, and thus will have different calendar intervals of follow-up. For purposes of evaluation, investigators will approach the VA-IHIE implementation as a patient-directed intervention given that additional information available from the exchange is available only on a patient-by-patient basis, i.e., a provider cannot use exchange information available for one patient in the care of another. Although the VA-IHIE program will be implemented at the site level, patients will be enrolled individually.

ELIGIBILITY:
Inclusion Criteria:

* Veteran's receiving care at the Indianapolis VAMC at least one year prior and one year post VA-IHIE enrollment
* Veteran's receiving care from a facility other than the Indianapolis VAMC one year prior and one year post VA-IHIE enrollment

Exclusion Criteria:

None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Veteran's receiving care at the Indianapolis VAMC
Sampling Method: Non-Probability Sample
Enrollment: 57073 (Actual)
Dates: Start 2012-12; Primary Completion 2015-06 (Actual); Study Completion 2016-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David A Haggstrom, MD, Principal Investigator — Richard L. Roudebush VA Medical Center, Indianapolis, IN
Locations (1):
- Richard L. Roudebush VA Medical Center, Indianapolis, IN, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Dixon BE, Haggstrom DA, Weiner M. Implications for informatics given expanding access to care for Veterans and other populations. J Am Med Inform Assoc. 2015 Jul;22(4):917-20. doi: 10.1093/jamia/ocv019. Epub 2015 Mar 31. PMID 25833394
- [Result] Kho AN, Cashy JP, Jackson KL, Pah AR, Goel S, Boehnke J, Humphries JE, Kominers SD, Hota BN, Sims SA, Malin BA, French DD, Walunas TL, Meltzer DO, Kaleba EO, Jones RC, Galanter WL. Design and implementation of a privacy preserving electronic health record linkage tool in Chicago. J Am Med Inform Assoc. 2015 Sep;22(5):1072-80. doi: 10.1093/jamia/ocv038. Epub 2015 Jun 23. PMID 26104741
- [Result] French DD, Margo CE, Campbell RR. Enhancing postmarketing surveillance: continuing challenges. Br J Clin Pharmacol. 2015 Oct;80(4):615-7. doi: 10.1111/bcp.12658. Epub 2015 Jun 1. No abstract available. PMID 25869078
- [Result] Byrne C, Hunolt E, Bouhaddou O, Pan E, Botts NE, Mercincavage L, Olinger L, Banty K, Bennett J, Weiner M, Haggstrom DA, Cromwell T. Performance evaluation framework for the Virtual Lifetime Electronic Record (VLER) health information exchange pilot program. AMIA ... Annual Symposium proceedings / AMIA Symposium. AMIA Symposium. 2013 Nov 16; 1(1):162.
- [Result] Dixon BE, Miller T, Overhage JM. Barriers to achieving the last mile in health information exchange: A survey of small hospitals and physician practices. Jounal of Healthcare Information Management. 2013 Oct 3; 27(4):53-58.
- [Result] French DD, Dixon BE, Perkins SM, Myers LJ, Weiner M, Zillich AJ, Haggstrom DA. Short-Term Medical Costs of a VHA Health Information Exchange: A CHEERS-Compliant Article. Medicine (Baltimore). 2016 Jan;95(2):e2481. doi: 10.1097/MD.0000000000002481. PMID 26765453
- [Result] Dixon BE, Ofner S, Perkins SM, Myers LJ, Rosenman MB, Zillich AJ, French DD, Weiner M, Haggstrom DA. Which veterans enroll in a VA health information exchange program? J Am Med Inform Assoc. 2017 Jan;24(1):96-105. doi: 10.1093/jamia/ocw058. Epub 2016 Jun 6. PMID 27274014
- [Result] Dixon BE, Barboza K, Jensen AE, Bennett KJ, Sherman SE, Schwartz MD. Measuring Practicing Clinicians' Information Literacy. An Exploratory Analysis in the Context of Panel Management. Appl Clin Inform. 2017 Feb 15;8(1):149-161. doi: 10.4338/ACI-2016-06-RA-0083. PMID 28197620
- [Result] Nguyen KA, Haggstrom DA, Ofner S, Perkins SM, French DD, Myers LJ, Rosenman M, Weiner M, Dixon BE, Zillich AJ. Medication Use among Veterans across Health Care Systems. Appl Clin Inform. 2017 Mar 8;8(1):235-249. doi: 10.4338/ACI-2016-10-RA-0184. PMID 28271121

RESULTS

PARTICIPANT FLOW:
Groups:
- Controls in Study (Not Enrolled in Health Care Exchange): Patients in this arm will represent Veterans seen at the Indianapolis VA Medical Center (VAMC) for whom information exchange has not been activated.
- Patients Enrolled in HIE: Patients in this arm will represent Veterans seen at the Indianapolis VAMC for whom information exchange has been activated by the patient choosing to "opt-in."
Period: Overall Study
Arm/Group | Controls in Study (Not Enrolled in Health Care Exchange) | Patients Enrolled in HIE
Started | 50446 | 6627
Completed | 50446 | 6627
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Baseline cohort consists of Veterans who had 2 outpatient, or 1 inpatient visit to the Indianapolis VAMC in the year prior to the index date of 3/1/12.
Groups:
- Controls in Study (Not Enrolled in Health Care Exchange): Patients in this arm will represent Veterans seen at the Indianapolis VAMC for whom information exchange has not been activated.
- Enrolled in HIE: Patients in this arm will represent Veterans seen at the Indianapolis VAMC for whom information exchange has been activated by the patient choosing to "opt-in."
- Total: Total of all reporting groups
Arm/Group | Controls in Study (Not Enrolled in Health Care Exchange) | Enrolled in HIE | Total
Number analyzed (Participants) | 50446 | 6627 | 57073
Age, Continuous [Median (Standard Deviation); unit: years] | 60.74 (15.77) | 62.17 (13.98) | 60.91 (15.58)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3607 | 514 | 4121
  Male | 46839 | 6113 | 52952
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 50446 | 6627 | 57073
Charlson Score [Median (Standard Deviation); unit: units on a scale] — Charlson comorbidity index is a scoring system which assigns points to varied conditions in an effort to determine severity of medical comorbidities. It is an integer scale with a theoretical range of 0 to 43. A score of 0 would represent a healthy individual with no significant comorbidities. A score of 3 would indicate an individual with significant number of comorbidities. An individual with a score of 8 would have several sever comorbidities. Any score above 8 would be unlikely as with that many comorbidities and individual would be incapacitated.
  units on a scale | .66 (1.42) | 1.25 (1.92) | .73 (1.5)

OUTCOME MEASURES:

1. Primary Outcome: Understanding Utilization of Healthcare Procedures by Veterans According to Source of Data
Description: Determining rates of usage of healthcare by veterans by source of data. This will clue us into any differences in utilization patterns between groups.
Time Frame: 2 years
Population: Veterans divided into enrolled and non-enrolled in HIE groups
Measure: Number; unit: participants
Groups:
- Controls in Study (Not Enrolled in Health Care Exchange): Patients in this group were not enrolled in Health Information Exchange.
- Enrolled in HIE: This group represents veterans were enrolled in Health Information Exchange via VLER
Arm/Group | Controls in Study (Not Enrolled in Health Care Exchange) | Enrolled in HIE
Number analyzed (Participants) | 50446 | 6627
participants
  VA Data Only | 41982 | 5073
  Data in Both Sources | 8358 | 1497
  Data only in Outside Source | 20 | 37
  No Data | 86 | 20

2. Primary Outcome: Effect of Health Information Exchange on Cost
Description: Before after analysis of the presence of health information exchange on costs within the VA healthcare system; Measure is cost, unadjusted, in dollars for the year post enrollment in the health information exchange
Time Frame: 2 Years
Population: 5269 individuals were excluded due to lacking cost information.
Measure: Median (Standard Deviation); unit: $ per year unadjusted total VA cost
Groups:
- Controls in Study (Not Enrolled in Health Care Exchange): Patients in this arm represent Veterans seen at the Indianapolis VAMC NOT enrolled in VLER who have readily identifiable cost information. The analysis will determine any difference among baseline variables
- Enrolled in HIE: Patients in this arm represent Veterans seen at the Indianapolis VAMC enrolled in VLER who have readily identifiable cost information. The analysis will determine any difference among baseline variables
Arm/Group | Controls in Study (Not Enrolled in Health Care Exchange) | Enrolled in HIE
Number analyzed (Participants) | 45700 | 6104
$ per year unadjusted total VA cost | 6,529 (9,153) | 9,915 (12,386)

3. Primary Outcome: Health Care Quality: Affect of HIE on LDL Levels of Participants.
Description: This study will measure the impact of HIE upon health care quality the underuse of ambulatory care services for diabetics. Measurements of underuse before and after implementation will detect improvements in the quality of care. To measure underuse, the study employs a measurement set that is sensitive to the potential effects and feasible for electronic data capture. In this specific instance, we expect the LDL levels to reflect lower numbers among diabetics due to greater health management via information sharing.
Time Frame: 3 years
Population: These are diabetics within the cohort defined as being diagnosed, alive, and being aged 18-75. Specifically looking at LDL
Measure: Least Squares Mean (95% Confidence Interval); unit: mg/dL of LDL
Groups:
- Control Prior to Intervention: Subjects not exposed to HIE prior to intervention
- Enrolled Prior to Intervention: Subjects enrolled in HIE prior to intervention
- Controls Post Intervention: Not enrolled in HIE post intervention
- Enrolled Post Intervention: Those participating in HIE post intervention
Arm/Group | Control Prior to Intervention | Enrolled Prior to Intervention | Controls Post Intervention | Enrolled Post Intervention
Number analyzed (Participants) | 1445 | 338 | 1445 | 338
mg/dL of LDL | 86.308 [85.677 to 86.938] | 85.263 [83.762 to 86.763] | 83.957 [83.321 to 84.592] | 82.640 [81.12 to 84.155]

4. Secondary Outcome: Health Care Quality: Care Sensitive Admissions
Description: This study will use the Agency for Healthcare Research and Quality's (AHRQ) Prevention Quality Indicators (PQI) to calculate the outcome measure. The PQIs are a set of measures used with hospital inpatient data to identify ambulatory care sensitive conditions. The PQIs consist of 14 conditions. The study will adopt 12 that are commonly used for adult patients: angina, asthma, bacterial pneumonia, chronic obstructive pulmonary disease, congestive heart failure, dehydration, diabetes long-term complications, diabetes short-term complications, diabetes uncontrolled, hypertension, lower-limb amputation among diabetes patients, and urinary infection.
Time Frame: 3 years
Population: This analysis looked specifically at hospitalizations within a cohort of diabetes patients (a subset of the whole).
Measure: Number; unit: ACS Hospitalizations per 100k patients
Groups:
- Pre-Intervention Control: Control subjects prior to intervention.
- Pre-Intervention Cases: Intervention subject prior to intervention
- Post-Intervention Control: Control subjects after intervention.
- Post -Intervention Cases: Intervention subject after intervention
Arm/Group | Pre-Intervention Control | Pre-Intervention Cases | Post-Intervention Control | Post -Intervention Cases
Number analyzed (Participants) | 11176 | 2149 | 11176 | 2149
ACS Hospitalizations per 100k patients | 2083 | 3229 | 2194 | 3350

ADVERSE EVENTS:
Description: As a retrospective data analysis, the possibility of adverse events caused by research affecting participating veterans was minimal. Steps were taken to prevent accidental disclosure of data as the key preventive effort in preventing adverse events.
Arm/Group | Controls in Study (Not Enrolled in Health Care Exchange) | Patients Enrolled in HIE
Serious Adverse Events (participants affected / at risk) | 0/50446 | 0/6627
Other Adverse Events (participants affected / at risk) | 0/50446 | 0/6627

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes